CLINICAL TRIAL: NCT04120207
Title: An Eight-week Randomised Controlled Trial of Home-based Pilates for Symptoms of Anxiety, Depression, and Fatigue Among People With MS With Minimal-to-mild Mobility Disability: Study Protocol
Brief Title: An Eight-week RCT of Home-based Pilates for Symptoms of Anxiety, Depression, and Fatigue Among People With MS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Limerick (Other)
Responsible Party: Principal Investigator, Karl Fleming, Structured PhD Student, University of Limerick
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: #2017_03_17_EHS
Record Dates: First submitted 2019-10-07; First posted 2019-10-09 (Actual); Last update posted 2019-10-09 (Actual); Status verified 2019-10

CONDITIONS: Multiple Sclerosis
Keywords: Pilates; Home-based; Anxiety; Depression; Fatigue
MeSH Terms: conditions — Multiple Sclerosis; Anxiety Disorders; Depression; Fatigue

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: The principal investigator was blinded to participant allocation, and the analyses were performed blinded to the group. Participants' individual identification numbers assigned at baseline were used during the course of the trial. Following full data extraction from SurveyMonkey.com, identifying information were removed, such that no participant could be identified in the working dataset through one, or a combination of different variables.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home-based Pilates (Experimental): This group will perform two weekly sessions of Pilates for eight weeks, completed with at least 48-hours between sessions, in their own home, supported by a DVD developed and previously implemented and evaluated by the lead researcher in a feasibility trial among people with Multiple Sclerosis. Each Pilates session will last approximately one hour and is comprised of seven Pilates warm-up exercises and fourteen mat-based beginner's level exercise. Four repetitions of each Pilates movement will be performed during sessions in the first two weeks, with intensity being self-regulated by the participant based on level of physical condition. Repetitions will gradually progress at biweekly intervals, resulting in ten repetitions being performed for the final two weeks of the trial (Weeks 7 and 8). Six post-training stretches will be maintained for a minimum of thirty seconds.
  Interventions: Behavioral: Home-based Pilates
- Delayed-Start Control (Other): Participants randomized to Delayed-start will be instructed to maintain their pre-intervention physical activity levels during the trial and will be contacted by the lead researcher by email or telephone to ensure timely completion of the on-line outcome assessments at biweekly intervals. Following the 8-week intervention, Delayed start participants will be provided with the Pilates DVD for their own use, but no data will be collected. For both groups, participants who experience a relapse will be immediately withdrawn from the study, which will be recorded by the lead researcher.
  Interventions: Other: Delayed-start Pilates

INTERVENTIONS:
Behavioral: Home-based Pilates — The Home-based Pilates group will complete two Pilates classes at home, twice weekly, for a period of eight weeks.
  Arms: Home-based Pilates
Other: Delayed-start Pilates — The Delayed-start group will maintain their regular daily activities, and be provided with a copy of the Pilates DVD following the intervention, for their own use.
  Arms: Delayed-Start Control

SUMMARY:
This study will investigate the effects of eight-weeks home-based Pilates on symptoms of anxiety, depression, and fatigue among people with Multiple Sclerosis. Half of participants will perform two weekly home-based Pilates sessions guided by a DVD, while the other half will maintain their regular daily activities.

DETAILED DESCRIPTION:
This will be a home-based, single blind, randomised, controlled trial comparing immediate-start home-based Pilates with a delayed-start control group. The study protocol was approved by the University Research Ethics Committee. Participants will provide written informed consent prior to testing. The home-based setting promotes national recruitment of participants through the MS Society of Ireland, via distribution of posters and participation information leaflets on social media and text alerts to members. Interested participants will be invited to contact the lead researcher via phone or email, who will answer any study-related questions. Potential participants will be screened for selection criteria over the phone and provided with Participant Information Sheet (PIS), informed consent, Physical Activity Readiness Questionnaire (PAR-Q), and Patient Determined Disease Steps (PDDS) form via post or email. Following screening and initial baseline testing, eligible participants will be randomized to immediate-start home-based Pilates, or delayed-start control, by an independent researcher who will not be involved in outcome assessments, using a computer-generated randomisation tool (www.randomizer.org). The Home-based Pilates group will perform two weekly sessions for eight weeks, completed with at least 48-hours between sessions, in their own home, supported by a DVD developed and previously implemented and evaluated by the lead researcher in a feasibility trial among people with Multiple Sclerosis. The instructor on the DVD is a certified Pilates Instructor. Each participant will receive documented details of the Pilates protocol, along with the DVD which will operate on a DVD player or participant's laptop computer. On activating the DVD, participants will be provided with an opening screen, offering four options to choose from; "Play all" plays the entire contents of the DVD from start to finish; "Warm Up", provides introductory teaching points on the core principles of Pilates along with teaching and demonstration of the Pilates' warm-up exercises; "Main Phase" provides demonstrations and key teaching points of the fourteen Pilates exercise routine, and "Post Stretch" demonstrates and teaches the post-stretch exercises. Each Pilates session will last approximately one hour and is comprised of seven Pilates warm-up exercises and fourteen mat-based beginner's level exercise. Four repetitions of each Pilates movement will be performed during sessions in the first two weeks, with intensity being self-regulated by the participant based on level of physical condition. Repetitions will gradually progress at biweekly intervals, resulting in ten repetitions being performed for the final two weeks of the trial (Weeks 7 and 8). Six post-training stretches will be maintained for a minimum of thirty seconds. Fidelity, adherence, dose and compliance shall be monitored via self-report exercise diaries containing session date, number of repetitions completed per exercise, and session RPE (Rate of perceived exertion), recorded by the participant immediately following session completion. Exercise diaries will be supplemented by a weekly telephone call consisting of direct questions about the frequency, intensity, and duration of the Pilates they have completed and whether they have experienced difficulties with exercise completion, any adverse events or relapses.

The Delayed-Start Control group be instructed to maintain their pre-intervention physical activity levels during the trial and will be contacted by the lead researcher by email or telephone to ensure timely completion of the on-line outcome assessments at biweekly intervals. Following the 8-week intervention, Delayed-Start participants will be provided with the Pilates DVD for their own use, but no data will be collected. For both groups, participants who experience a relapse will be immediately withdrawn from the study, which will be recorded by the lead researcher.

ELIGIBILITY:
Inclusion Criteria: Adults with self-reported, physician-diagnosed Multiple Sclerosis PDDS score <3 Free from any other significant physical or psychiatric condition Have no previous Pilates experience

-

Exclusion Criteria: Have any medical contraindications to safe participation in physical activity established by the PAR-Q

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-08-28 (Actual); Study Completion 2019-08-28 (Actual)

PRIMARY OUTCOMES:
Profile of Mood States - Brief Form (POMS-B) | Baseline
  The 30-item POMS-B assesses the intensity of feelings of tension, depressed mood, energy and fatigue. Participants respond to each item "based on how you feel RIGHT NOW" using a 5-point Likert scale ranging from 0 (not at all) to 4 (Extremely). Each subscale score ranges from 0-20. The psychometric properties of the POMS-B are well established.
Profile of Mood States - Brief Form (POMS-B) | Week 2
  The 30-item POMS-B assesses the intensity of feelings of tension, depressed mood, energy and fatigue. Participants respond to each item "based on how you feel RIGHT NOW" using a 5-point Likert scale ranging from 0 (not at all) to 4 (Extremely). Each subscale score ranges from 0-20. The psychometric properties of the POMS-B are well established.
Profile of Mood States - Brief Form (POMS-B) | Week 4
  The 30-item POMS-B assesses the intensity of feelings of tension, depressed mood, energy and fatigue. Participants respond to each item "based on how you feel RIGHT NOW" using a 5-point Likert scale ranging from 0 (not at all) to 4 (Extremely). Each subscale score ranges from 0-20. The psychometric properties of the POMS-B are well established.
Profile of Mood States - Brief Form (POMS-B) | Week 6
  The 30-item POMS-B assesses the intensity of feelings of tension, depressed mood, energy and fatigue. Participants respond to each item "based on how you feel RIGHT NOW" using a 5-point Likert scale ranging from 0 (not at all) to 4 (Extremely). Each subscale score ranges from 0-20. The psychometric properties of the POMS-B are well established.
Profile of Mood States - Brief Form (POMS-B) | Week 8
  The 30-item POMS-B assesses the intensity of feelings of tension, depressed mood, energy and fatigue. Participants respond to each item "based on how you feel RIGHT NOW" using a 5-point Likert scale ranging from 0 (not at all) to 4 (Extremely). Each subscale score ranges from 0-20. The psychometric properties of the POMS-B are well established.
State Trait Anxiety Inventory (STAI-Y1) | Baseline
  The 20-item State and Trait subscales of the widely used and well-validated STAI will assess anxiety. Participants rate each item using a 4-point Likert scale, from 1 "Not at all" to 4 "Very much so". Total score ranges from 20-80; higher scores indicate greater anxiety. The STAI has well-documented psychometric properties in people with MS.
State Trait Anxiety Inventory (STAI-Y1) | Week 2
  The 20-item State and Trait subscales of the widely used and well-validated STAI will assess anxiety. Participants rate each item using a 4-point Likert scale, from 1 "Not at all" to 4 "Very much so". Total score ranges from 20-80; higher scores indicate greater anxiety. The STAI has well-documented psychometric properties in people with MS.
State Trait Anxiety Inventory (STAI-Y1) | Week 4
  The 20-item State and Trait subscales of the widely used and well-validated STAI will assess anxiety. Participants rate each item using a 4-point Likert scale, from 1 "Not at all" to 4 "Very much so". Total score ranges from 20-80; higher scores indicate greater anxiety. The STAI has well-documented psychometric properties in people with MS.
State Trait Anxiety Inventory (STAI-Y1) | Week 6
  The 20-item State and Trait subscales of the widely used and well-validated STAI will assess anxiety. Participants rate each item using a 4-point Likert scale, from 1 "Not at all" to 4 "Very much so". Total score ranges from 20-80; higher scores indicate greater anxiety. The STAI has well-documented psychometric properties in people with MS.
State Trait Anxiety Inventory (STAI-Y1) | Week 8
  The 20-item State and Trait subscales of the widely used and well-validated STAI will assess anxiety. Participants rate each item using a 4-point Likert scale, from 1 "Not at all" to 4 "Very much so". Total score ranges from 20-80; higher scores indicate greater anxiety. The STAI has well-documented psychometric properties in people with MS.
Hospital Anxiety and Depression Scale (HADS) | Baseline
  The 7-item anxiety and depression subscales of the 14-item HADS measures anxiety and depressive symptoms in the prior week. Subscale scores range from 0-21 with higher scores indicative of greater anxiety and depressive symptoms, and validated cut-scores ≥8 classify anxiety and depression caseness. The HADS has demonstrated reasonable psychometric properties among people with Multiple Sclerosis, demonstrating acceptable sensitivity (90% and 89% for the depression subscale) and specificity (87% and 81% for the anxiety subscale).
Hospital Anxiety and Depression Scale (HADS) | Week 2
  The 7-item anxiety and depression subscales of the 14-item HADS measures anxiety and depressive symptoms in the prior week. Subscale scores range from 0-21 with higher scores indicative of greater anxiety and depressive symptoms, and validated cut-scores ≥8 classify anxiety and depression caseness. The HADS has demonstrated reasonable psychometric properties among people with Multiple Sclerosis, demonstrating acceptable sensitivity (90% and 89% for the depression subscale) and specificity (87% and 81% for the anxiety subscale).
Hospital Anxiety and Depression Scale (HADS) | Week 4
  The 7-item anxiety and depression subscales of the 14-item HADS measures anxiety and depressive symptoms in the prior week. Subscale scores range from 0-21 with higher scores indicative of greater anxiety and depressive symptoms, and validated cut-scores ≥8 classify anxiety and depression caseness. The HADS has demonstrated reasonable psychometric properties among people with Multiple Sclerosis, demonstrating acceptable sensitivity (90% and 89% for the depression subscale) and specificity (87% and 81% for the anxiety subscale).
Hospital Anxiety and Depression Scale (HADS) | Week 6
  The 7-item anxiety and depression subscales of the 14-item HADS measures anxiety and depressive symptoms in the prior week. Subscale scores range from 0-21 with higher scores indicative of greater anxiety and depressive symptoms, and validated cut-scores ≥8 classify anxiety and depression caseness. The HADS has demonstrated reasonable psychometric properties among people with Multiple Sclerosis, demonstrating acceptable sensitivity (90% and 89% for the depression subscale) and specificity (87% and 81% for the anxiety subscale).
Hospital Anxiety and Depression Scale (HADS) | Week 8
  The 7-item anxiety and depression subscales of the 14-item HADS measures anxiety and depressive symptoms in the prior week. Subscale scores range from 0-21 with higher scores indicative of greater anxiety and depressive symptoms, and validated cut-scores ≥8 classify anxiety and depression caseness. The HADS has demonstrated reasonable psychometric properties among people with Multiple Sclerosis, demonstrating acceptable sensitivity (90% and 89% for the depression subscale) and specificity (87% and 81% for the anxiety subscale).
Quick Inventory of Depressive Symptomatology (QIDS) | Baseline
  The 16-item QIDS will assess depressive symptom severity across nine core criteria for depression, based on the prior week. Participants will rate severity and frequency of specific symptoms experienced in the prior week. Total scores range from 0-27, with a higher score illustrating more symptom severity. Scores >5 indicate at least mild depression. The QIDS is a valid measure to quantify depressive symptoms with good sensitivity and specificity among people with Multiple Sclerosis.
Quick Inventory of Depressive Symptomatology (QIDS) | Week 2
  The 16-item QIDS will assess depressive symptom severity across nine core criteria for depression, based on the prior week. Participants will rate severity and frequency of specific symptoms experienced in the prior week. Total scores range from 0-27, with a higher score illustrating more symptom severity. Scores >5 indicate at least mild depression. The QIDS is a valid measure to quantify depressive symptoms with good sensitivity and specificity among people with Multiple Sclerosis.
Quick Inventory of Depressive Symptomatology (QIDS) | Week 4
  The 16-item QIDS will assess depressive symptom severity across nine core criteria for depression, based on the prior week. Participants will rate severity and frequency of specific symptoms experienced in the prior week. Total scores range from 0-27, with a higher score illustrating more symptom severity. Scores >5 indicate at least mild depression. The QIDS is a valid measure to quantify depressive symptoms with good sensitivity and specificity among people with Multiple Sclerosis.
Quick Inventory of Depressive Symptomatology (QIDS) | Week 6
  The 16-item QIDS will assess depressive symptom severity across nine core criteria for depression, based on the prior week. Participants will rate severity and frequency of specific symptoms experienced in the prior week. Total scores range from 0-27, with a higher score illustrating more symptom severity. Scores >5 indicate at least mild depression. The QIDS is a valid measure to quantify depressive symptoms with good sensitivity and specificity among people with Multiple Sclerosis.
Quick Inventory of Depressive Symptomatology (QIDS) | Week 8
  The 16-item QIDS will assess depressive symptom severity across nine core criteria for depression, based on the prior week. Participants will rate severity and frequency of specific symptoms experienced in the prior week. Total scores range from 0-27, with a higher score illustrating more symptom severity. Scores >5 indicate at least mild depression. The QIDS is a valid measure to quantify depressive symptoms with good sensitivity and specificity among people with Multiple Sclerosis.
Modified Fatigue Impact Scale (MFIS) | Baseline
  The 21-item MFIS is a recommended core outcome measure in exercise studies in people with Multiple Sclerosis, that measures physical, cognitive and psychosocial components of fatigue. Participants respond to "how often fatigue has affected you in this way during the past 4 weeks", using a 5-point Likert scale ranging from 0 (Never) to 4 (Almost Always). Physical subscale scores range from 0 to 36, Cognitive from 0 to 40, and Psychosocial from 0 to 8. Total MFIS scores (0 to 84), is computed by summing physical, cognitive, and psychosocial subscale scores, with a higher score indicating greater impact of fatigue on participant activities. A total fatigue cut-off score of ≥38 distinguishes between fatigued and non-fatigued individual. It has been proposed by the Multiple Sclerosis Council for Clinical Practice Guidelines as a reliable assessment tool of perceived fatigue (1998), with excellent test-retest reliability, and good correlation with the Fatigue Severity Scale.
Modified Fatigue Impact Scale (MFIS) | Week 2
  The 21-item MFIS is a recommended core outcome measure in exercise studies in people with Multiple Sclerosis, that measures physical, cognitive and psychosocial components of fatigue. Participants respond to "how often fatigue has affected you in this way during the past 4 weeks", using a 5-point Likert scale ranging from 0 (Never) to 4 (Almost Always). Physical subscale scores range from 0 to 36, Cognitive from 0 to 40, and Psychosocial from 0 to 8. Total MFIS scores (0 to 84), is computed by summing physical, cognitive, and psychosocial subscale scores, with a higher score indicating greater impact of fatigue on participant activities. A total fatigue cut-off score of ≥38 distinguishes between fatigued and non-fatigued individual. It has been proposed by the Multiple Sclerosis Council for Clinical Practice Guidelines as a reliable assessment tool of perceived fatigue (1998), with excellent test-retest reliability, and good correlation with the Fatigue Severity Scale.
Modified Fatigue Impact Scale (MFIS) | Week 4
  The 21-item MFIS is a recommended core outcome measure in exercise studies in people with Multiple Sclerosis, that measures physical, cognitive and psychosocial components of fatigue. Participants respond to "how often fatigue has affected you in this way during the past 4 weeks", using a 5-point Likert scale ranging from 0 (Never) to 4 (Almost Always). Physical subscale scores range from 0 to 36, Cognitive from 0 to 40, and Psychosocial from 0 to 8. Total MFIS scores (0 to 84), is computed by summing physical, cognitive, and psychosocial subscale scores, with a higher score indicating greater impact of fatigue on participant activities. A total fatigue cut-off score of ≥38 distinguishes between fatigued and non-fatigued individual. It has been proposed by the Multiple Sclerosis Council for Clinical Practice Guidelines as a reliable assessment tool of perceived fatigue (1998), with excellent test-retest reliability, and good correlation with the Fatigue Severity Scale.
Modified Fatigue Impact Scale (MFIS) | Week 6
  The 21-item MFIS is a recommended core outcome measure in exercise studies in people with Multiple Sclerosis, that measures physical, cognitive and psychosocial components of fatigue. Participants respond to "how often fatigue has affected you in this way during the past 4 weeks", using a 5-point Likert scale ranging from 0 (Never) to 4 (Almost Always). Physical subscale scores range from 0 to 36, Cognitive from 0 to 40, and Psychosocial from 0 to 8. Total MFIS scores (0 to 84), is computed by summing physical, cognitive, and psychosocial subscale scores, with a higher score indicating greater impact of fatigue on participant activities. A total fatigue cut-off score of ≥38 distinguishes between fatigued and non-fatigued individual. It has been proposed by the Multiple Sclerosis Council for Clinical Practice Guidelines as a reliable assessment tool of perceived fatigue (1998), with excellent test-retest reliability, and good correlation with the Fatigue Severity Scale.
Modified Fatigue Impact Scale (MFIS) | Week 8
  The 21-item MFIS is a recommended core outcome measure in exercise studies in people with Multiple Sclerosis, that measures physical, cognitive and psychosocial components of fatigue. Participants respond to "how often fatigue has affected you in this way during the past 4 weeks", using a 5-point Likert scale ranging from 0 (Never) to 4 (Almost Always). Physical subscale scores range from 0 to 36, Cognitive from 0 to 40, and Psychosocial from 0 to 8. Total MFIS scores (0 to 84), is computed by summing physical, cognitive, and psychosocial subscale scores, with a higher score indicating greater impact of fatigue on participant activities. A total fatigue cut-off score of ≥38 distinguishes between fatigued and non-fatigued individual. It has been proposed by the Multiple Sclerosis Council for Clinical Practice Guidelines as a reliable assessment tool of perceived fatigue (1998), with excellent test-retest reliability, and good correlation with the Fatigue Severity Scale.

SECONDARY OUTCOMES:
Seven-day Physical Activity Recall Scale (7d-PAR) | Baseline
  This measures the approximate number of hours the subject slept and how much time they engaged in moderate, hard, and very hard activity. It is a valid measure used extensively in MS research, and has demonstrated high test-retest reliability.
Seven-day Physical Activity Recall Scale (7d-PAR) | Week 2
  This measures the approximate number of hours the subject slept and how much time they engaged in moderate, hard, and very hard activity. It is a valid measure used extensively in MS research, and has demonstrated high test-retest reliability.
Seven-day Physical Activity Recall Scale (7d-PAR) | Week 4
  This measures the approximate number of hours the subject slept and how much time they engaged in moderate, hard, and very hard activity. It is a valid measure used extensively in MS research, and has demonstrated high test-retest reliability.
Seven-day Physical Activity Recall Scale (7d-PAR) | Week 6
  This measures the approximate number of hours the subject slept and how much time they engaged in moderate, hard, and very hard activity. It is a valid measure used extensively in MS research, and has demonstrated high test-retest reliability.
Seven-day Physical Activity Recall Scale (7d-PAR) | Week 8
  This measures the approximate number of hours the subject slept and how much time they engaged in moderate, hard, and very hard activity. It is a valid measure used extensively in MS research, and has demonstrated high test-retest reliability.
Godin Leisure-Time Exercise Questionnaire (GLTEQ) | Baseline
  This is a self-report measure of physical activity in persons with multiple sclerosis. Its validity is well established in MS, and it is sensitive to change following active interventions. Frequency of strenuous (e.g., running or jogging), moderate (e.g., fast walking, easy swimming), and mild (e.g., easy walking) exercise performed for more than 15 minutes during leisure time over a usual week was recorded. Total weekly leisure activity scores were calculated as follows, (strenuous x 9) + (moderate x 5) + (mild x 3). Scores (>=24) indicate activity levels to provide substantial benefits towards overall health contribution.
Godin Leisure-Time Exercise Questionnaire (GLTEQ) | Week 2
  This is a self-report measure of physical activity in persons with multiple sclerosis. Its validity is well established in MS, and it is sensitive to change following active interventions. Frequency of strenuous (e.g., running or jogging), moderate (e.g., fast walking, easy swimming), and mild (e.g., easy walking) exercise performed for more than 15 minutes during leisure time over a usual week was recorded. Total weekly leisure activity scores were calculated as follows, (strenuous x 9) + (moderate x 5) + (mild x 3). Scores (>=24) indicate activity levels to provide substantial benefits towards overall health contribution.
Godin Leisure-Time Exercise Questionnaire (GLTEQ) | Week 4
  This is a self-report measure of physical activity in persons with multiple sclerosis. Its validity is well established in MS, and it is sensitive to change following active interventions. Frequency of strenuous (e.g., running or jogging), moderate (e.g., fast walking, easy swimming), and mild (e.g., easy walking) exercise performed for more than 15 minutes during leisure time over a usual week was recorded. Total weekly leisure activity scores were calculated as follows, (strenuous x 9) + (moderate x 5) + (mild x 3). Scores (>=24) indicate activity levels to provide substantial benefits towards overall health contribution.
Godin Leisure-Time Exercise Questionnaire (GLTEQ) | Week 6
  This is a self-report measure of physical activity in persons with multiple sclerosis. Its validity is well established in MS, and it is sensitive to change following active interventions. Frequency of strenuous (e.g., running or jogging), moderate (e.g., fast walking, easy swimming), and mild (e.g., easy walking) exercise performed for more than 15 minutes during leisure time over a usual week was recorded. Total weekly leisure activity scores were calculated as follows, (strenuous x 9) + (moderate x 5) + (mild x 3). Scores (>=24) indicate activity levels to provide substantial benefits towards overall health contribution.
Godin Leisure-Time Exercise Questionnaire (GLTEQ) | Week 8
  This is a self-report measure of physical activity in persons with multiple sclerosis. Its validity is well established in MS, and it is sensitive to change following active interventions. Frequency of strenuous (e.g., running or jogging), moderate (e.g., fast walking, easy swimming), and mild (e.g., easy walking) exercise performed for more than 15 minutes during leisure time over a usual week was recorded. Total weekly leisure activity scores were calculated as follows, (strenuous x 9) + (moderate x 5) + (mild x 3). Scores (>=24) indicate activity levels to provide substantial benefits towards overall health contribution.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew P Herring, PhD, Principal Investigator — University of Limerick
Locations (1):
- University of Limerick, Limerick, Ireland

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Primary outcome data will be made available for five years at six months following publication of primary outcome summary data. Secondary outcome data will be made available for five years at six months following publications of secondary outcome summary data.
Access Criteria: Requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Derived] Fleming KM, Coote SB, Herring MP. Home-based Pilates for symptoms of anxiety, depression and fatigue among persons with multiple sclerosis: An 8-week randomized controlled trial. Mult Scler. 2021 Dec;27(14):2267-2279. doi: 10.1177/13524585211009216. Epub 2021 Apr 19. PMID 33870785